CLINICAL TRIAL: NCT02159092
Title: The Role of Contingency Management in Waterpipe Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington State University (Other)
Responsible Party: Principal Investigator, kawkab shishani, Assistant Professor, Washington State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5K01DA037661-02 (NIH)
Record Dates: First submitted 2014-06-05; First posted 2014-06-09 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Waterpipe Smoking
Keywords: Waterpipe; Smoking cessation; Contingency management; Dependence
MeSH Terms: conditions — Water Pipe Smoking; Smoking Cessation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Contingency Management (Experimental): Monetary incentives are given for submitting negative saliva cotinine tests.
  Interventions: Behavioral: Contingency Management
- Fixed Rate Control (No Intervention): Fixed amounts of payments are provided for submitting saliva samples

INTERVENTIONS:
Behavioral: Contingency Management — Monetary incentive for the CM groups is contingent on a saliva cotinine reading that indicates smoking abstinence. Participants were assessed 10 times (Mondays/Thursdays) for abstinence from smoking waterpipe verified by saliva cotinine. The maximum monetary incentives this group can receive is $192.50. The CM groups followed an escalating schedule where: 1) the dollar amount of the incentive increases by $.50 as long as the participant is abstinent at each visit;; and 2) resets to the starting incentive ($14) if the participant was non-compliant at the previous visit, but is compliant at the current visit. Also, Participants were given $10 bonus for every three consecutive compliant visits.
  Arms: Contingency Management

SUMMARY:
Tobacco use kills more than 500,000 people in the United States each year. Although the use of cigarettes has declined, the use of other tobacco products has remained steady. Waterpipe smoking is a common form of tobacco smoking after cigarettes in the U.S. In fact, in 2007 the American Lung Association issued a policy alert to warn consumers about this first new tobacco trend of the 21st century (American Lung Association, 2007). Few studies have been conducted on waterpipe smoking to investigate its harmful effects. Furthermore, no known studies have evaluated treatments for smoking cessation in waterpipe smokers. This study aims to test the role of contingency management (CM) in promoting abstinence from waterpipe smoking for 5 weeks verified by salivary cotinine and to characterize self-reported nicotine withdrawal symptoms. Based on the alarming growth rate over a short period of time in waterpipe tobacco smoking, there is a critical need for clinical research to investigate treatment modalities targeting smoking cessation for waterpipe smokers. Given the evidence for the role of CM in promoting abstinence from many types of drug use, investigation of the utility of CM for waterpipe smoking cessation is important and timely. Although Nicotine Replacement Therapy is the mainstay treatment for treating nicotine dependence delivered through cigarettes, the intermittent use patterns that characterize waterpipe smoking suggest that CM may be more effective in promoting waterpipe smoking cessation. The evidence based knowledge generated in this study may assist in the translation of the treatment program into public health practice.

DETAILED DESCRIPTION:
Contingency Management (CM) has been used successfully to treat tobacco addiction. CM is a powerful drug abuse treatment modality for facilitating change in drug use behaviors. The utility of CM as a treatment for waterpipe smoking is logical, but needs to be evaluated as a tool in the treatment of waterpipe smoking. The primary objective of this research plan is to test the role of CM in promoting abstinence from waterpipe tobacco smoking. The specific aims of the research include: specific aim 1: Conduct a feasibility study to test if CM promotes abstinence from nicotine delivered through waterpipe; specific aim 2: Characterize self-reported nicotine withdrawal symptoms. A randomized clinical trial involving eligible participants who are randomly assigned with equal allocation to either Contingency Management (CM) or Fixed Rate Control (FRC) will be conducted. A 2-group (CM versus FRC) x 10 (repeated measures) mixed-model design will be used. Participants in this study will be followed for 5 weeks during which smoking abstinence will be measured 10 times. Reinforcement in the form of monetary payment delivered contingent on the participant's salivary cotinine will be provided

ELIGIBILITY:
Inclusion Criteria:

* Must be18 years and older
* Smoked waterpipe average of >12 times per month for 2 years

Exclusion Criteria:

* Smokes cigarettes (self-report)
* Uses any tobacco product (self-report)
* Uses illicit drugs (urine analysis for toxicology)
* Interested in quitting waterpipe smoking (self-report)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
quitting waterpipe smoking | 5 weeks
  Quitting waterpipe smoking will be assessed using saliva cotinine test twice a week for five weeks. Also, participants will be asked at each visit if they have smoked waterpipe during the past days between visits.

SECONDARY OUTCOMES:
withdrawal symptoms | 5 weeks
  Withdrawal symptoms will be assessed using the Minnesota Withdrawal Scale-Revised (MNWS-R) and the Questionnaire of Smoking Urges (QSU). These self-report measures will be completed twice a week for five weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Kawkab Shishani, PhD, Principal Investigator — Washington State University
Locations (1):
- South Campus Facility, Washington State University, Spokane, Washington, United States